CLINICAL TRIAL: NCT05632185
Title: Equine-assisted Therapy Effectiveness in Improving Emotion Regulation, Self-efficacy, and Perceived Self-esteem of Patients Suffering From Substance Use Disorder
Brief Title: Equine-assisted Therapy Effectiveness in Improving Emotion Regulation of Patients Suffering From Substance Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMBSUREC/06112022
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2022-11

CONDITIONS: Substance Use Disorder (SUD)
MeSH Terms: conditions — Substance-Related Disorders | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: one group will receive Equine assisted intervention, and a control group to receive the regular care used in the setting
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): standard regular treatment modalities
- Equine assisted intervention (Active Comparator): patients will receive weekly equine-assisted therapy sessions over a period of 8 weeks in addition to their standard regular therapy
  Interventions: Behavioral: Equine-assisted Therapy

INTERVENTIONS:
Behavioral: Equine-assisted Therapy — An equine therapy session typically consists of specific tasks and challenges to overcome, with the aid and guidance of horses. There is no riding involved and no specific skills are necessary to take part in these sessions
  Arms: Equine assisted intervention

SUMMARY:
Substance Use Disorder (SUD) is a term replacing the diagnoses of abuse and dependence adopted in DSM-4 and DSM-5 . It is an overwhelming public health problem throughout the world, with increasing trends throughout the last few decades. This study aims to assess the effectiveness of quine-assisted addiction therapy in improving emotion regulation, self-efficacy, and perceived self-esteem among patients suffering from substance use disorders. This open-label randomized controlled trial study will be conducted at Behman hospital, Helwan, Cairo, Egypt.

It will include all patients suffering substance use disorder randomized into two equal groups: one group will receive Equine assisted intervention, and a control group to receive the regular care used in the setting. A self-administered questionnaire with tools for emotion regulation questionnaire, General Self-efficacy (GSE) scale, and Self- Esteem will be used to collect data.

DETAILED DESCRIPTION:
Research design: A randomized controlled trial design will be utilized in this study.

Setting: The study will conduct Behman hospital, Helwan, Cairo, Egypt. It was founded in 1940 as the first private psychiatric hospital in Egypt. With a 210-bed capacity, the hospital is considered as one of the biggest medical centers in Helwan, Egypt. The hospital is the pioneer of equine psychotherapy in Egypt.

Duration of the Study: The four phases of data collection are expected to take 6 months, from December 2022 to May 2023.

Subjects: The study population will consist of all Patients suffering from substance use disorder receiving their care at Behman hospital, during the time of the study. The inclusion criteria will be being adult diagnosed with substance use disorder, hospitalized for at least one month in the study hospital, and physically able to deal with horses. Those patients suffering from any other physical or psychological ailments preventing them from active participation in the intervention will exclude. The remaining patients will equally randomized, using simple random numbers computer program, into an intervention group to receive the equine assisted therapy and a control group to receive the regular care used in the setting.

Data collection tools: Data will be collected using a self-administered questionnaire with standardized tools for assessment of emotion regulation, General Self-Efficacy, and perceived self-esteem, in addition to a section for the demographic and disease characteristics developed by the researchers. This cover data about patient age, gender, current marital status, place of residence, educational level, current job status, income, as well as age at start and duration of substance of use etc.

The first tool emotion regulation questionnaire developed by Gross and John (2003). It will be used to assess how respondents tend to regulate their emotions positively through cognitive reappraisal, or negatively through expressive suppression. It consists of ten statements: 6 for cognitive reappraisal (such as "When I want to feel more positive emotion, I change the way I'm thinking about the situation"), and 4 for expressive suppression (4 statements such as "When I am feeling negative emotions, I make sure not to express them"). The responses are on a 7-point Likert-type scale ranging from "strongly disagree" to "strongly agree." The scores of each dimension are summed giving a maximum total score of 42 for the appraisal dimension and 28 for the suppression dimension. A higher score indicates more appraisal or more suppression. Scoring is kept continuous according to tool instructions. The tool demonstrated high validity and reliability in previous studies (Mauss et al., 2005; Ochsner and Gross, 2005).

The second tool will be the General Self-efficacy (GSE) scale developed by Schwarzer and Jerusalem (1995). It also has 10 statements on a 4-point Likert type scale ranging from "not at all true" (scored 1) to "exactly true" (scored 4). Examples of statements are: "It is easy for me to stick to my aims and accomplish my goals," and "I can solve most problems if I invest the necessary effort." A total score ranging from 10 to 40 is obtained simple summation of items' scores. A higher score denotes more GSE. The reliability of the tool as well as its concurrent and predictive validity were documented (Schwarzer and Jerusalem, 2010).

The third tool will be the self-esteem test developed by Sorensen (2006). The tool has 50 statements such as: "I often feel like I don't know what is expected of me," and "I am not vey aware of my feelings." The respondent is asked to check the statements he/she feels true for him/her. The number of items checked is calculated, ranging from zero to 50. A higher number indicates lower self-esteem. The tool was validated and showed good reliability (Martín-Albo et al., 2007).

ELIGIBILITY:
Inclusion Criteria:

adult diagnosed with substance use disorder, hospitalized for at least one month in the study hospital, and physically able to deal with horses

Exclusion Criteria:

other physical or psychological ailments preventing them from active participation in the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
emotion regulation questionnaire | Six months
  assess how respondents tend to regulate their emotions positively through cognitive reappraisal, or negatively through expressive suppression.
General Self-efficacy (GSE) scale | Six months
  10 statements on a 4-point Likert type scale ranging from "not at all true" (scored 1) to "exactly true" (scored 4)
the self-esteem test | Six months
  50 statements such as: "I often feel like I don't know what is expected of me," and "I am not vey aware of my feelings." The respondent is asked to check the statements he/she feels true for him/her.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Souilm, Doctor, Principal Investigator — Bani-Suef University
Locations (1):
- Behman hospital, Helwan, Cairo, Egypt, Cairo, Egypt